CLINICAL TRIAL: NCT03762590
Title: GENetic Education Risk Assessment and TEsting Study (GENERATE)
Brief Title: GENetic Education Risk Assessment and TEsting Study
Acronym: GENERATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Mayo Clinic (Other); M.D. Anderson Cancer Center (Other); Johns Hopkins University (Other); University of California, San Diego (Other); Weill Medical College of Cornell University (Other); Stand Up To Cancer (Other); Lustgarten Foundation (Other)
Responsible Party: Principal Investigator, Sapna Syngal, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-222
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Candidates for Hereditary Pancreatic Cancer Testing
Keywords: Candidates for Hereditary Pancreatic Cancer Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxy.me plus Color Genomics Arm (Arm 1) (Experimental): * Participants in this arm will receive genetic education through an online platform called Doxy.me
  * The Doxy.me session will consist of two parts: 1) a pre-recorded genetic education video 2) a live interactive video conferencing session with a GENERATE genetic counselor
  * After completing the Doxy.me session and post intervention questionnaires, participants will be directed to the Color Genomics study portal where they may elect to review Color Genomics' genetic education content or proceed directly to order genetic testing
  * Intervention is Doxy.me genetic education +/- genetic education via Color Genomics website
  Interventions: Other: Doxy.me genetic education +/- Color Genomics genetic education
- Color Genomics Only Arm (Arm 2) (Experimental): * Participants in this arm will access genetic education on the Color Genomics website which includes both written information and an educational video
  * After accessing the Color Genomics website, participants may elect to review educational content or proceed directly to order genetic testing
  * Intervention is genetic education via Color Genomics website
  Interventions: Other: Color Genomics genetic education

INTERVENTIONS:
Other: Doxy.me genetic education +/- Color Genomics genetic education — Doxy.me is a HIPAA compliant telemedicine platform that allows clinicians to provide education to remote patients.
  Genetic education via Doxy.me will consist of a pre-recorded genetic education video and a live interactive video conferencing session with a GENERATE genetic counselor.
  Genetic education via Color Genomics will consist of both written information and an educational video on the Color Genomics website.
  Arms: Doxy.me plus Color Genomics Arm (Arm 1)
Other: Color Genomics genetic education — Genetic education via Color Genomics will consist of both written information and an educational video on the Color Genomics website.
  Arms: Color Genomics Only Arm (Arm 2)

SUMMARY:
The goal of the GENERATE Study is to improve genetic testing and cancer prevention in family members of pancreatic cancer patients who may have genetic mutations (inherited changes). The study will measure how different methods of genetic education increase the rate of genetic testing in these families.

This is an investigational study to measure the effects of two methods of genetic education. Participants may elect to undergo genetic testing as part of the study and will be asked to provide a saliva sample via a saliva-testing kit. The genetic testing done in this study is FDA approved and will be processed in a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory.

Up to 1,000 participants will be enrolled in this study.

DETAILED DESCRIPTION:
Around 1 in 10 (10%) pancreatic cancer patients carries an inherited change (mutation) in a gene which can increase the risk of cancer. Relatives of patients with pancreatic cancer are often unaware that the mutation can be passed down through the family. Having information about genetic risk can be important to family members. There may be options for early and/or more frequent screening (to look for cancer or pre-cancer) or early detection recommendations.

This research is being done to study the impact of different methods of teaching about and offering genetic testing to family members of pancreatic cancer patients who may carry a mutation.

Study arms:

Individuals will be randomized (like flipping a coin) by family to one of the two study arms to receive genetic education and elect to undergo genetic testing.

Individuals in Arm 1 (video conference platform plus Color Genomics) will receive genetic education via a pre-recorded educational video and interactive session with the study team through an internet-based platform.

Individuals in Arm 2 (Color Genomics Only) will receive genetic education from Color Genomics, Inc., an online, commercial genetic testing service.

Informed consent:

Participants will be asked to provide informed consent in order to join the study.

Study questionnaires:

Questionnaires will be given at baseline and throughout the duration of the study. Participants will be asked to complete questionnaires through the online study database, called REDCap (paper questionnaires are also an option). The baseline questionnaires will ask participants about their medical history, their experience with pancreatic cancer and other relevant health behaviors.

The follow-up questionnaires will ask about how much participants worried about cancer, how participants made choices, their knowledge gained and how much families shared genetic test results (if participants chose to get testing). The study will also ask about participants' choices to have pancreas exams and other surveillance (long-term screening) procedures, and their lifestyle choices after receiving the intervention.

Genetic testing:

GENERATE offers genetic testing at no cost to participants in the study. Color Genomics will provide the genetic testing services for the study. Participants will be directed to create a personal Color Genomics account that will allow them to enter their personal and family history information, keep track of their genetic testing kit and receive their genetic test results. Participants will be mailed an FDA-approved saliva collection kit from Color Genomics. When participants receive the kit in the mail, they will be able to use the kit's unique barcode number to activate it and link it to their online account. A video on the website will show participants how to provide a large enough saliva sample. It will also contain instructions for how to properly package and mail back the kit to Color Genomics using a pre-paid shipping package.

Getting test results:

It usually takes about 4-6 weeks to get the results back from this genetic test. Participants will receive an email letting them know that their results are available for review through their Color Genomics account or via a phone call with a Color Genomics genetic counselor.

Length of study:

The total participation on this study will last about 18 months, including follow-up. Participants may be contacted regarding participation in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Individual who is 18 years or older
* Individual who has signed the informed consent
* Individual with:

  --A first-degree relative who has (or had) pancreatic ductal adenocarcinoma (PDAC) OR a second-degree relative who has (or had) PDAC and has a known germline mutation in APC, ATM, BRCA1, BRCA2, CDKN2A, EPCAM, MLH1, MSH2, MSH6, PALB2, PMS2, STK11, or TP53
* The germline mutation and history of PDAC must be on the maternal side or paternal side of the individual's family
* Individual with a valid United States mailing address
* Individual with access to a healthcare provider and is willing to share genetic test results with that provider/the study team

Exclusion Criteria:

* Individual with a known cancer susceptibility gene
* Individual who has received genetic counseling for cancer risk within the last 3 years
* Individual who has received a bone marrow transplant, who has had a blood transfusion within the last 7 days, or who has an active hematologic malignancy (i.e. leukemia or lymphoma)
* Individual who is unable to sign the informed consent because of mental incompetency or psychiatric illness
* Individual who is unwilling to complete baseline and follow-up questionnaires
* Individual who has a life expectancy of less than 1 year
* Individual with only APC I1307K mutation within their family
* Individual with only PMS2 exons 12-15 deletion mutation within their family

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of genetic testing among family members of mutation positive PDAC patients, among family members of mutation positive individuals with a family history of PDAC and among first-degree relatives of PDAC patients | 2 years
  Measure the effect that alternative methods of genetic education and delivery models have on the increase of genetic testing among family members of mutation positive PDAC patients, among family members of mutation positive individuals with a family history of PDAC and among first-degree relatives of PDAC patients in each arm of the intervention study. We will document how many relatives per family elect to undergo genetic testing and compare the results of this measure between both arms of the study.

SECONDARY OUTCOMES:
Level of cancer-risk distress | Baseline, immediately post intervention, 3-4 months post intervention, 15 months post intervention
  Measure the degree that individuals worry about getting cancer using the adapted Lerman Breast Cancer Worry Scale. This is an 8 item scale with a total score ranging from 8-32, with high scores indicating more frequent worries. A cut-off of equal to or greater than 14 will indicate moderate to high cancer worry.
Increase of knowledge of genetic testing | Immediately post intervention
  Assess the participants' understanding of general concepts learned within a genetic counseling session targeted towards multigene panel testing, including inheritance, inherited cancer risks, possible test results of multi-gene panel testing and limitations, and changes in medical management related to an inherited cancer risk
Factors in decision making | Immediately post intervention
  Assess the participants perception of how helpful the genetic education was in deciding to pursue genetic testing using a validated 10 item Preparation for Decision Making Scale. This is a brief validated 10 item measure that assesses the participants perception of how useful a decision support intervention is in preparing the participant to make a health decision. Items are summed and scored, and higher scores indicate higher perceived level of preparation.
Degree of family communication about genetic test results | 3-4 months post intervention, 15 months post intervention
  Measure items pertaining to disclosure of genetic test results to relatives which includes asking if participants communicated at all with specific family members and if they disclosed results of genetic testing to anyone in their family
Uptake of surveillance for pancreatic, other associated cancers and health behaviors | Baseline and 15 months post intervention
  Examine appropriate screening (such as mammography, colonoscopy) uptake and health behaviors (i.e. smoking, alcohol use) for those who test positive or negative in both arms of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Syngal, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.

REFERENCES:
- [Derived] Rodriguez NJ, Furniss CS, Yurgelun MB, Ukaegbu C, Constantinou PE, Fortes I, Caruso A, Schwartz AN, Stopfer JE, Underhill-Blazey M, Kenner B, Nelson SH, Okumura S, Zhou AY, Coffin TB, Uno H, Horiguchi M, Ocean AJ, McAllister F, Lowy AM, Klein AP, Madlensky L, Petersen GM, Garber JE, Lippman SM, Goggins MG, Maitra A, Syngal S. A Randomized Trial of Two Remote Health Care Delivery Models on the Uptake of Genetic Testing and Impact on Patient-Reported Psychological Outcomes in Families With Pancreatic Cancer: The Genetic Education, Risk Assessment, and Testing (GENERATE) Study. Gastroenterology. 2024 May;166(5):872-885.e2. doi: 10.1053/j.gastro.2024.01.042. Epub 2024 Feb 5. PMID 38320723